CLINICAL TRIAL: NCT01194791
Title: A Multicentric, Phase II Trial of Lenalidomide, Cyclophosphamide and Dexamethasone in Patients With Primary Systemic Amyloidosis (AL) Newly Diagnosed, Not Candidates for Hematopoietic Stem Cell Transplantation
Brief Title: Lendexal in Patients With Primary Systemic Amyloidosis (AL) Newly Diagnosed
Acronym: LENDEXAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENDEXAL; 2009-017707-28 (EudraCT Number)
Record Dates: First submitted 2010-07-26; First posted 2010-09-03 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2015-11

CONDITIONS: Primary Systemic Amyloidosis
Keywords: Amyloidosis; Lenalidomide
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Lenalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, Cyclophosphamide and Dexamenthasone (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 15 mg by mouth for 21 days followed by 7 days rest during 6 cycles
  Other Names: Lendexal
Drug: Cyclophosphamide — Cyclophosphamide 300 mg/m2, on days 1 and 8 every 4 weeks during 6 cycles
Drug: Dexamethasone — Oral dexamethasone 20 mg/day on days 1-4 and 9-12 given at 4-week intervals during 6 cycles

SUMMARY:
Primary outcome measure:

- Hematologic response rate to the association of Lenalidomide, Cyclophosphamide and Dexamethasone.

Secondary outcome measures:

* Organ response rate.
* Predictors of response (cardiac biomarkers, serum free light chains).
* Toxicity
* Safety (type, frequency, severity and relationship of adverse events to the study drug).
* Duration of response.
* Time to progression.
* Overall survival

DETAILED DESCRIPTION:
It is a multicenter, single arm treatment, phase II study of the combination in one treatment arm with Lenalidomide, Cyclophosphamide and Dexamethasone.

Subjects who qualify for participation will receive lenalidomide plus dexamethasone and cyclophosphamide in 4-week cycles. Subjects will be seen (study visits) every 2 weeks for the first 3 cycles of therapy and monthly thereafter.

Cycles of lenalidomide/dexamethasone/cyclophosphamide will consists of lenalidomide 15 mg by mouth for 21 days followed by 7 days rest and 300 mg/m2 of cyclophosphamide on days 1 and 8 plus oral dexamethasone 20 mg/day on days 1-4 and 9-12 given at 4-week intervals. Patients will be treated with 6 cycles of therapy with the option to continue beyond as long there is evidence of response. In this case the dose of lenalidomide will be the same and the dose of the dexamethasone will be administered only on days 1 to 4 of each cycle and the dose of cyclophosphamide only day 1 during 6 cycles. After 12 cycles if the patients remaining in response, will be treated with 10 mg/day, cyclophosphamide day 1, and dexamethasone will be administered on days 1 to 4 of each cycle.

For the first 3 cycles, patients will be followed for adverse events with hematologic control every 2 weeks and monthly thereafter. Patients will be required to have a blood work-up including total serum protein and serum protein electrophoresis, urine protein studies and a clinical visit before each cycle. Organ involvement will be assessed every 4 cycles during the first year of therapy. Hematologic response will be assessed every 3 months and organ response every 6 months after the first year of treatment.

Treatment modifications will be based on adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE Version 3.0).

There will be 30 patients enrolled.

The trial consists of three periods: pre-treatment, treatment and follow up period.

Pre-treatment phase: include the enrolment visit in order to determine if the patient is eligible to participate in the study. The patient will sign the Informed Consent Form to take part in the study, and will receive detailed information about the treatment, its benefits and risks.

Treatment phase: include the 12 cycles of 28 days treatment with Lenalidomide, Cyclophosphamide and Dexamethasone as induction therapy followed with low doses of Lenalidomide and Dexamethasone during three years until progression or unacceptable toxicity levels.

Follow up phase: Once the clinical trial has finished, patients will be followed during usual clinical practice visits where progression, free survival and overall survival will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age > 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements according with investigator criteria.
* Diagnosis of symptomatic primary systemic amyloidosis based on tissue Congo red positive staining as well as positive immunohistochemical staining for light chains or presence of a monoclonal protein in serum and/or urine or clonal bone marrow plasma cells
* Previously untreated disease
* Patients should not candidates for up-front high-dose therapy/stem cell transplantation
* Serologically measurable disease defined as follows:

Evidence of a monoclonal light chain in serum and urine by immunofixation Raise of the level of circulating free light chains above the ordinary limits and an abnormal relationship kappa/lambda.

* Performance status ECOG ≤ 2 (see Annex 3).
* Laboratory tests results within these ranges:

Absolute neutrophil count ≥ 1 x 10 9/ L. Platelet count ≥ 100 x 10 9/ L Serum creatinine less than 3.0 mg/dL Serum bilirubin less than 3.0 mg/dL

- Females of childbearing potential (FCBP) must agree to: Know the teratogenic risks of the study drug

Commit to use contraceptives during the 4 weeks before the start of this study drug treatment, during the treatment and also 4 weeks after it, even amenorrheic cases. All of it applies always except women committed to maintain sexual abstinence confirming it monthly. Some of effective contraceptives are:

Birth control implant Levonorgestrel-releasing intrauterine device. Depot medroxyprogesterone acetate Tubal ligation Sexual intercourse only with a vasectomized partner. The effectiveness of vasectomy must be confirmed by two semen analysis; the result must be negative Inhibiting ovulation pill progesterone only (for example: desogestrel) if it is determined that the patient doesn't use an effective contraceptive method will be referred to a skilled health professional to receive advice on contraception, so that they can begin to birth control measures.

It's discouraged combine oral contraceptives in myeloma multiple women cases treated with Lenalidomide combined with Dexamethasone due to high venous thromboembolism risk. In case these kind of patient were having combined oral contraceptives, she must change to another one of list above. Risks of venous thromboembolism will remain during the 3 or 4 weeks after discontinue combine oral contraceptives treatment. Concomitant treatment with dexamethasone reduces the effectiveness of contraceptive steroids.

Implants and levonorgestrel-releasing intrauterine systems are related to higher risks of infections at the moment of the implant or when there is metrorrhagia. It should be considered prophylactic treatment with antibiotics for neutropenic patients.

Normally it's discouraged copper intrauterine devices because of the infection risk and menstrual blood loss at the moment of the implant for patients with neutropenia or thrombocytopenia.

Women patients must follow all warnings for an effective contraception, even if she is amenorrheic.

Women patients must be aware about effects of pregnancy and go to a health care centre urgently in case of pregnancy risk.

She must take a pregnancy test with a minimum sensitivity of 25 mUl/ml, under medical supervision, when the study visits or three days before the visit, when she were 4 weeks at least using effective contraceptive methods. This requirement applies for women who practice a complete and continuous sexual abstinence. Test should confirm that the patient is not pregnant at the time of starting treatment.

She must take a pregnancy test, under medical supervision, each 4 weeks, even a pregnancy test 4 weeks after the end of the study treatment, except in case of a confirmed tubal ligation. Pregnancy test should be performed the day of the study's visit or during the three days before it. This requirement also applies for childbearing women who practice a complete and continuous sexual abstinence.

- Male patients must: Undertake to use latex condoms during treatment with study medication including all periods of interruption of doses, even one week after finishing treatment if his partner is a woman of childbearing who doesn't use contraceptive methods.

Commit not to donate semen during treatment with study medication and even one week after finishing treatment.

- All patients should: Refrain from donating blood during treatment with study medication and even one week after finishing treatment.

Refrain from sharing the study medication with other people and return unused study medication to the investigator or the pharmacist.

Exclusion Criteria:

* Localized cutaneous AL, only carpal tunnel syndrome, merely vascular amyloid in the bone marrow biopsy, AL in a plasmacytoma or AL associated to multiple myeloma (>30% plasma cells in bone marrow, lytic bone lesions, hypercalcemia, plasmacytomas).
* Other causes of amyloidosis (secondary, familial, senile).
* Candidates for high dose chemotherapy/ stem cell transplant.
* Previously treated AL.
* Any condition including laboratory abnormalities, which placed the subjects at unacceptable risk if he/she were to participating the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days prior to baseline.
* Any prior use of lenalidomide
* Any cancer in the previous 5 years, except no melanoma skin cancer, cervix or prostate cancer treated in the initial state with prostate-specific antigen within normal limits.
* Known positive for HIV.
* Cardiac ejection fraction below 50%
* Pregnant or breast-feeding (can not breast-feed while taking lenalidomide)
* Patients who are not able to use antithrombotic prophylaxis or reject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hematologic response rate to the association of Lenalidomide, Cyclophosphamide and Dexamethasone | 6 months

SECONDARY OUTCOMES:
Organ response rate | 6 months
Predictors of response (cardiac biomarkers, serum free light chains) | 5 years
Safety and tolerability | 5 years
Duration of response | 10 years
Time to progression | 5 years
Overall survival | 10 yeras

CONTACTS AND LOCATIONS:
Overall Officials: Bladé Joan, Dr, Study Chair — Hospital Clinic of Barcelona
Locations (10):
- Spain (10):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Morales Messeguer, Murcia
  - Hospitalm Clínico de Salamanca, Salamanca
  - Hospital La Fe, Valencia
  - Hospital Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Cibeira MT, Oriol A, Lahuerta JJ, Mateos MV, de la Rubia J, Hernandez MT, Granell M, Fernandez de Larrea C, San Miguel JF, Blade J; PETHEMA cooperative study group. A phase II trial of lenalidomide, dexamethasone and cyclophosphamide for newly diagnosed patients with systemic immunoglobulin light chain amyloidosis. Br J Haematol. 2015 Sep;170(6):804-13. doi: 10.1111/bjh.13500. Epub 2015 May 14. PMID 25974382
- See also: Spanish Haematology Association — http://aehh.org
- See also: CRO — http://seif88.com